CLINICAL TRIAL: NCT04614818
Title: A Multi-center, Retrospective Analysis of Clinical Character, Outcome and Prognosis of Lymphoepithelioma-like Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Tongyu Lin, Professor, Sun Yat-sen University
Other Study IDs: B2020-289-01
Record Dates: First submitted 2020-10-26; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Lymphoepithelioma-Like Carcinoma; Lymphoepithelioma-Like Carcinoma of Thymus; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- pulmonary lymphoepithelioma-like carcinoma: The primary site of lymphoepithelioma-like carcinoma locates in the lungs.
  Interventions: Other: Non-intervention research
- lymphoepithelioma-like carcinoma of thymus: The primary site of lymphoepithelioma-like carcinoma locates in the thymus.
  Interventions: Other: Non-intervention research
- lymphoepithelioma-like carcinoma of salivary glands: The primary site of lymphoepithelioma-like carcinoma locates in the parotid gland or submandibular gland.
  Interventions: Other: Non-intervention research
- lymphoepithelioma-like carcinoma of stomach: The primary site of lymphoepithelioma-like carcinoma locates in the stomach.
  Interventions: Other: Non-intervention research
- lymphoepithelioma-like carcinoma of esophagus: The primary site of lymphoepithelioma-like carcinoma locates in the esophagus.
  Interventions: Other: Non-intervention research
- lymphoepithelioma-like carcinoma of liver: The primary site of lymphoepithelioma-like carcinoma locates in the liver.
  Interventions: Other: Non-intervention research
- lymphoepithelioma-like carcinoma of ovaries: The primary site of lymphoepithelioma-like carcinoma locates in the ovaries.
  Interventions: Other: Non-intervention research
- lymphoepithelioma-like carcinoma of cervix: The primary site of lymphoepithelioma-like carcinoma locates in the cervix.
  Interventions: Other: Non-intervention research
- lymphoepithelioma-like carcinoma of tonsil: The primary site of lymphoepithelioma-like carcinoma locates in the tonsil.
  Interventions: Other: Non-intervention research

INTERVENTIONS:
Other: Non-intervention research — Non-intervention research

SUMMARY:
The investigators retrospective collect the clinical data of patients diagnosed with lymphoepithelioma-like carcinoma, including primary site, gender, age, smoking history, tumor stage, time of initial treatment, EBV-DNA copy number, first-line treatment and survival status.

DETAILED DESCRIPTION:
Lymphoepithelioma-like carcinoma (LELC) is a rare EBV-related tumor. Its histology is similar to that of nasopharyngeal carcinoma. In 2004, the WHO classified LELC into one subtype of large cell carcinoma, and the 2015 WHO classified it as other and unclassified cancers. LELC can originate in many organs, including parotid glands, throat, lungs, digestive tract, genitourinary system, etc. Driver gene mutations are rarely seen, and most of them are PD-L1 positive. In terms of treatment, there is no standard first-line treatment for lymphoepithelioma-like cancer. Patients with early-stage lymphoepithelioma-like cancer can receive surgery or radiotherapy, while palliative radiotherapy or chemotherapy is the main treatment for patients in advanced stage. The survival time is about 107 months, the 5-year OS is 59.5%, which is better than the prognosis of lung squamous cell carcinoma in the same period. A retrospective study of Sun yat-sen University Cancer Hospital included 127 patients with advanced lung LELC who received first-line chemotherapy between 2007 and 2018. Gemcitabine and platinum based chemotherapy and paclitaxel and platinum based regimens are significantly better than pemetrexed and platinum, but most of the current studies on lymphoepithelioma-like cancer focus on LELC that originates in the lung. But for other sites, such as parotid glands, liver, digestive tract, are mostly based on case reports, and there are few retrospective studies with large samples to explore their clinical features and treatment outcome. Therefore, investigators designed this retrospective clinical study to analyze the clinical characteristics, treatment, survival, and prognostic risk factors of patients with lymphoepithelioma-like carcinoma in order to summary the clinical character and guide treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Lymphoepithelioma-like carcinoma confirmed by histopathology;
* 2. The primary lesion does not involve the nasopharynx;
* 3. Complete data for patient's character, laboratory and imaging test, treatment and follow-up are available.

Exclusion Criteria:

* 1. Concomitant with other tumor components at the time of diagnosis;
* 2. Have a history of any other malignant tumors;
* 3. Lack of complete data

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed diagnosis of lymphoepithelioma-like carcinoma of any primary site, including lung, salivary glands, thymus, tonsil, liver, stomach, esophagus, ovary, cervix et al.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of diagnosis until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.

SECONDARY OUTCOMES:
Overall survival | From date of diagnosis until the date of death from any cause, whichever came first, assessed up to 24 months.
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu Q, Wang W, Zhou P, Fu Y, Zhang Y, Shao YW, Jiang L. Primary pulmonary lymphoepithelioma-like carcinoma is characterized by high PD-L1 expression, but low tumor mutation burden. Pathol Res Pract. 2020 Aug;216(8):153043. doi: 10.1016/j.prp.2020.153043. Epub 2020 Jun 2. PMID 32703503
- [Background] Fang W, Hong S, Chen N, He X, Zhan J, Qin T, Zhou T, Hu Z, Ma Y, Zhao Y, Tian Y, Yang Y, Xue C, Tang Y, Huang Y, Zhao H, Zhang L. PD-L1 is remarkably over-expressed in EBV-associated pulmonary lymphoepithelioma-like carcinoma and related to poor disease-free survival. Oncotarget. 2015 Oct 20;6(32):33019-32. doi: 10.18632/oncotarget.5028. PMID 26361045
- [Background] He J, Shen J, Pan H, Huang J, Liang W, He J. Pulmonary lymphoepithelioma-like carcinoma: a Surveillance, Epidemiology, and End Results database analysis. J Thorac Dis. 2015 Dec;7(12):2330-8. doi: 10.3978/j.issn.2072-1439.2015.12.62. PMID 26793355
- [Background] Abouelfad DM, Yassen NN, Amin HAA, Shabana ME. Lymphoepithelioma-Like Carcinoma of the Breast Mimicking Granulomatous Mastitis- Case Report and Review of the Literature. Asian Pac J Cancer Prev. 2017 Jul 27;18(7):1737-1741. doi: 10.22034/APJCP.2017.18.7.1737. PMID 28749097
- [Derived] Chen M, Chen Y, Fang X, Wang Z, Pu X, Liang C, Guo H, Li Q, Pan F, Hong H, Huang H, Li J, Lin T. Clinical features and treatment outcome of lymphoepithelioma-like carcinoma from multiple primary sites: a population-based, multicentre, real-world study. BMC Pulm Med. 2022 Sep 22;22(1):360. doi: 10.1186/s12890-022-02097-6. PMID 36138362